CLINICAL TRIAL: NCT00653900
Title: Does Platelet Function Testing Help us Assess Intraoperative Bleeding Risk in Cardiac and Vascular Surgery for Patients Who Are on Plavix Prior to Admission?
Brief Title: Platelet Function Testing Help and Intraoperative Bleeding Risk for Patients Who Are on Plavix Prior to Surgery
Status: Withdrawn | Type: Observational
Why Stopped: insufficient funding
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Dr Suhail Dohad, PI, CSMC
Other Study IDs: Pro00013820
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Perioperative Bleeding
Keywords: Verify now; platelet function; platelet function testing; bleeding risk; periprocedural bleeding; clopidogrel; Our initial goal is to establish if a certain degree of; platelet function abnormality can predict a higher bleeding; or higher transfusions.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1 drop of blood for the "verify now" test, which is done before the procedure.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All patients undergoing elective, invasive cardiac procedure on plavix prior to admission

SUMMARY:
A large number of patients are currently on Antiplatelet inhibition using aspirin or Plavix therapy (A Thieno pyridine - ADP mediated platelet inhibitor). A group of these patients often require Cardiac and/or Vascular surgical procedures. These patients are at a higher risk for perioperative bleeding complications and higher re-operation/re-exploration for bleeding and subsequent blood product transfusions.

The aim of this protocol is to assess platelet function via the "Verify Now" device prior to surgery. The Verify Now device requires a small drop of fresh blood for each sample and is an FDA approved device.

The investigators initial goal is to establish if a certain degree of platelet function abnormality can predict a higher bleeding complication or higher transfusions (Phase I, 20 patients). This initial study will allow us to determine a sample size for Phase II. Phase II will maintain the same protocol, however after completion of Phase I, a more accurate sample size determination can be made. Additionally, the investigators want to establish if knowledge of platelet dysfunction will change procedure technique or preparation to lower bleeding and/or lead to cancellation/rescheduling of procedure (Phase III).

Participants will be those patients who are taking plavix and are undergoing vascular or cardiac surgery. They will undergo a platelet function evaluation measured as Platelet Response Unit (PRU) via the "verify now" device on admission/pre surgery. This test involves taking 1 drop of blood from the patient, one time, before the procedure. The Verify Now device is FDA approved.

Perioperative bleeding will be assessed by absolute drop in hematocrit immediate post-op compared to the immediate preoperative value. An additional discharge hematocrit will be used if no blood products have been used during the initial hospital stay. Hematocrit evaluation via a complete blood count is a part of standard patient care. Additionally, utilization of blood products (factors, PLT, PRBC's, etc.) will be assessed.

In order to conduct the research, patients will be identified by reviewing the OR schedule. All consecutive patients on ASA/Plavix will be mailed a letter in order to introduce them to the study. The letter provides a phone number to call if the patient does NOT want to receive a phone call from the investigative staff. This letter is uploaded under item 18-02 of the study application. If patients do not call the office, then the investigative staff will call the potential participants to introduce the study. Final consent will be completed in PACU on arrival at the hospital for planned surgical procedure.

A Hematocrit will be performed on the consented patient preoperatively, immediately post-op, and at discharge. A PRU will be assessed using a few drops of the patients' blood preoperatively (PACU). Patients' records will be reviewed to assess use of blood products. No additional follow up is required.

Patients' care will be no different than current standard of care, other than the 1 "verify now" test, which is done before the procedure.

ELIGIBILITY:
Inclusion Criteria:

* All consenting participants who are taking plavix prior to undergoing vascular or cardiac surgery.

Exclusion Criteria:

* All consenting participants who are NOT taking plavix prior to undergoing vascular or cardiac surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be those patients who are taking plavix and are undergoing vascular or cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06-03 (Actual); Study Completion 2009-06-03 (Actual)

PRIMARY OUTCOMES:
Perioperative bleeding (absolute drop in hematocrit, utilization of blood products (factors, PLT, PRBC's, etc.) will be assessed. | measured until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Suhail Dohad, MD, Principal Investigator — Attending Physician
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States